CLINICAL TRIAL: NCT00869453
Title: Gut Hormone Secretion Pattern in Response to Different Macronutrients in Healthy Volunteers
Brief Title: Gut Hormone Secretion and Macronutrients
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, professor of physiology, University of Lausanne
Other Study IDs: 162/08/CE/FBM
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Volunteers
Keywords: Gut hormone; hyperglycaemic clamp; glucose turnver
MeSH Terms: interventions — Glucose; CD36 Antigens; Proteins

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy volunteers
  Interventions: Other: test meal; Other: glucose; Other: fat; Other: protein; Other: control

INTERVENTIONS:
Other: test meal — Mixed meal containing bread, butter, beef
Other: glucose — administration of a glucose meal
Other: fat — administration of a lipid meal
Other: protein — administration of a protein meal
Other: control — no meal

SUMMARY:
The role of gut hormone (GLP-1, GIP, PYY...) in glucose homeostasis has been widely demonstrated. Furthermore modifications in their pattern of secretion seem to be involved in the improvement of glucose control in obese patients after bariatric surgery.

The purpose of this study is to assess the respective role of carbohydrate, fat and protein from a complete meal in gut hormones secretion.

DETAILED DESCRIPTION:
The study is designed to asses the role of each individual macronutrient of a compete meal in gut hormones secretion in healthy volunteers.

8 healthy young male subjects will be studied on 5 different occasions. To asses the role of each macronutient the subjects will recieve one of the following test meal: a complete sandwich, the proteic part of this complete meal, the glucidic part and the lipidic part. The fifth test will be a fasting test.

To assess the entero-insular axis, a 5.5 hours hyperglycaemic clamp will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-35 years old
* 19 kg/m2 ≤ BMI ≤ 25 kg/m2
* Healthy
* Low to moderate physical activity
* Non smokers

Exclusion Criteria:

* Family history of diabetes mellitus
* Any medication
* Participation to blood spending or other clinical study in the 3 months before the beginning of this study
* Consumption of drugs
* Consumption of more than 50g of alcool in a week
* Vegetarian or particular diet
* Anamnèse d'intolérance alimentaire
* Family history of food intolerance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Gut hormone secretion | within 4 hours following a test meal

SECONDARY OUTCOMES:
Entero-insular axis measurement | within 4 hours following a test meal
Glucose turnover | 6 hours
Insulin sensitivity | 6 hours
Substrate oxidation | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (2):
- Switzerland (2):
  - Cardiomet Clinical research Center, CHUV, Lausanne, Canton of Vaud
  - University of Lausanne, Lausanne

REFERENCES:
- [Derived] Carrel G, Egli L, Tran C, Schneiter P, Giusti V, D'Alessio D, Tappy L. Contributions of fat and protein to the incretin effect of a mixed meal. Am J Clin Nutr. 2011 Oct;94(4):997-1003. doi: 10.3945/ajcn.111.017574. Epub 2011 Aug 17. PMID 21849595